CLINICAL TRIAL: NCT02771860
Title: Randomized, Double Blind, Placebo-controlled Study to Evaluate the Efficacy of Denosumab 60mg sc Every 3 Months in Patients With Erosive Osteoarthritis of the Interphalangeal (IP) Finger Joints
Brief Title: RANKL-blockade for the Treatment of Erosive Osteoarthritis (OA) of Interphalangeal Finger Joints
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGO/2015/008; 2015-003223-53 (EudraCT Number)
Record Dates: First submitted 2016-03-18; First posted 2016-05-13 (Estimated); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-05

CONDITIONS: Hand Osteoarthritis
Keywords: denosumab; RANKL-blockade
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: denosumab (Active Comparator): 50 patients will be enrolled in this group for a total treatment duration of 24 months (96 weeks): 48 weeks denosumab 60mg sc every 12 weeks followed by a 48-weeks open label phase denosumab 60mg sc every 12 weeks. Calcium and vit D supplementation will be installed at baseline.
  Interventions: Drug: denosumab; Dietary Supplement: Calcium/Vit D supplementation
- Comparator (Placebo Comparator): 50 patients will be enrolled in this group for a total treatment duration of 24 months (96 weeks): 48 weeks placebo sc every 12 weeks followed by a 48-weeks open label phase denosumab 60mg sc every 12 weeks.
  Calcium and vit D supplementation will be installed at baseline
  Interventions: Drug: denosumab; Drug: Placebo; Dietary Supplement: Calcium/Vit D supplementation

INTERVENTIONS:
Drug: denosumab — 60mg sc
  Other Names: Active Comparator
Drug: Placebo — identical syringe
  Other Names: placebo comparator
  Arms: Comparator
Dietary Supplement: Calcium/Vit D supplementation — Daily dosage Calcium 1000mg / Vit D 880 IU
  Other Names: Steovit forte

SUMMARY:
This is a randomized, double blind placebo controlled one-site proof-of-concept study in subjects with erosive osteoarthritis (OA) of interphalangeal (IP) finger joints.

A total of 100 subjects will be enrolled into the study: 48 weeks placebo controlled double-blind phase with denosumab 60mg every 12 weeks, followed by a 48-week open-label phase in which all subjects will receive denosumab.

DETAILED DESCRIPTION:
Investigational therapy: denosumab 60mg subcutaneous injection every 12 weeks. All subjects will receive Calcium/vit D supplementation.

Efficacy objectives:

The primary objective is to assess the effect of denosumab on the reduction of radiographic erosive progression using the Ghent University Score System (GUSS).

The secondary objective is to assess the effect of denosumab on the reduction of radiographic erosive progression as defined by diminishing the appearance of new erosive IP finger joints.

The exploratory objective is mainly to assess the effect of denosumab on clinical variables, as well as ultrasonography and dual energy x-ray absorptiometry parameters.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects with hand OA having suffered from transient inflammatory attacks of the interphalangeal finger joints characteristic for what has been termed 'inflammatory' or 'erosive' hand OA.

  * Subjects with hand OA showing inflammatory signs, either clinically or ultrasonographically, of the interphalangeal finger joints.
  * Subjects with hand OA in which at least 1 interphalangeal finger joint has the typical appearance on the X-rays of a 'J' or 'E' phase joint as defined by the criteria mentioned above.
  * Subjects with hand OA where at least 1 interphalangeal finger joint in the 'J' or 'E' phase presents a palpable swelling.

Exclusion Criteria:

* Patients with known hypersensitivities to mammalian-derived drug preparations.
* Patients with clinically significant hypersensitivity to any of the components of Prolia.
* Current and/or Prior treatment with any investigational agent within 90 days, or five half-lives of the product, whichever is longer.
* Previous administration of denosumab from clinical trials or others (e.g. commercial use).
* Vitamin D deficiency [25(OH) vitamin D level < 20 ng/mL (< 49.9 nmol/L)]. Possibility of replenishment and re-screening.
* Subjects with current hypo- or hypercalcemia (normal serum calcium levels: 8.5-10.5 mg/dl or 2.12-2.62 mmol/L).
* Patients currently under bisphosphonate (BP) treatment or any use of oral BPs within 12 months of study enrollment or intravenous BPs or strontium ranelate within 5 years of study enrollment
* Prior use of any chondroprotective drug within 90 days e.g. chondroitin sulfate, glucosamine, avocado-soybean unsaponifiables, tetracyclins, corticosteroids.
* Prior use of any immunomodulating drug with possible effects on proinflammatory cytokine metabolism within 90 days a.o. corticosteroids, methotrexate, sulfasalazine, leflunomide, D-Penicillin, anti-malarials, cytotoxic drugs, tumor necrosis factor (TNF) blocking agents.
* History of drug or alcohol abuse in the last year.
* Patients suffering from chronic inflammatory rheumatic disease (e.g. rheumatoid arthritis, spondylarthropathy, psoriatic arthritis, gout, chondrocalcinosis or other auto-immune diseases, e.g. systemic lupus erythematosus).
* History of cancer or lymphoproliferative disease other than a successfully and completely treated squamous cell or basal cell carcinoma of the skin or cervical dysplasia, with no recurrence within the last two years.
* History of any Solid Organ or Bone Marrow Transplant.
* Comorbidities: significant renal function impairment (glomerular filtration < 30 ml/min/1.73m2 or <50% of normal value), uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure (NYHA III, IV), uncontrolled hypo or hyperparathyroidism, active inflammatory bowel disease, malabsorption, liver failure or chronic hepatic disease (serum aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) levels 3 times above normal), recent stroke (within three months), chronic leg ulcer and any other condition (e.g,. indwelling urinary catheter) which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures .
* Patient who is pregnant or planning pregnancy; if the female subject is of child-bearing age, she must use a valid mean of contraception during the study and for 9 months after last dose of study medication. For males with a partner of childbearing potential: subject refuses to use 1 effective methods of contraception for the duration of the study and for 10 months after the last dose of study medication.
* Female subjects who are breast-feeding.
* History of osteonecrosis of the jaw, and/or recent (within 3 months) tooth extraction or other unhealed dental surgery; or planned invasive dental work during the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Elewaut, Prof. Dr., Principal Investigator — UZ Ghent; August Verbruggen, Prof Dr. Em., Principal Investigator — UZ Ghent; Ruth Wittoek, Prof. Dr., Principal Investigator — UZ Ghent
Locations (1):
- UZ Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Experimental: Denosumab: 51 patients were enrolled in this group for a total treatment duration of 24 months (96 weeks): 48 weeks denosumab 60mg sc every 12 weeks followed by a 48-weeks open label phase denosumab 60mg sc every 12 weeks.
- Comparator - Placebo: 49 patients were enrolled in this group for a total treatment duration of 24 months (96 weeks): 48 weeks placebo sc every 12 weeks followed by a 48-weeks open label phase denosumab 60mg sc every 12 weeks.
Period: Overall Study
Arm/Group | Active Comparator: Experimental: Denosumab | Comparator - Placebo
Started | 51 | 49
Completed | 46 | 46
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Experimental: Denosumab | Comparator - Placebo | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 40 | 82
  >=65 years | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (7.7) | 60.6 (7.9) | 61.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 37 | 78
  Male | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 51 | 49 | 100
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m²] | 25.3 (3.5) | 25.3 (4.0) | 25.3 (3.8)
Number of radiographically affected joints [Mean (Standard Deviation); unit: count] — Any radiographically defined S, J, E, R joint, according to the Verbruggen and Veys score of 16 joints per patient
  count | 3.6 (2.2) | 4.0 (2.2) | 3.8 (2.2)
Ghent University scoring system (GUSS) of all joints [Mean (Standard Deviation); unit: units on a scale] — The Ghent University Scoring System, GUSS, is quantitative radiographic scoring system and found to be a reliable method to score radiographic change over time in erosive IP OA. It includes assessment of proportions of normal subchondral bone, subchondral plate and joint space over time. Range of score: min: 0 max:300. Change scores are measured where positive changes corresponds with remodeling or repair (better outcome), and negative changes with erosive progression (worse outcome).
  All joints refer to all proximal and distal IP joints (n = 16) (excluding 1st IP) in a patient.
  units on a scale | 249 (66) | 248 (67) | 249 (67)
Ghent University scoring system (GUSS) of target joints [Mean (Standard Deviation); unit: units on a scale] — The Ghent University Scoring System, GUSS, is quantitative radiographic scoring system and found to be a reliable method to score radiographic change over time in erosive IP OA. It includes assessment of proportions of normal subchondral bone, subchondral plate and joint space over time. Range of score: min: 0 max:300. Change scores are measured where positive changes corresponds with remodeling or repair (better outcome), and negative changes with erosive progression (worse outcome).
  Target joints are predefined at baseline according to the protocol.
  units on a scale | 155.9 (69.3) | 158.7 (46.8) | 157.3 (58.3)
Pain [Mean (Standard Deviation); unit: units on a scale] — on a numerical rating scale (0-10), with 0 corresponds to no pain and 10 to maximal pain
  units on a scale | 4.7 (2.5) | 4.8 (2.7) | 4.8 (2.7)
Australian-Canadian Hand Osteoarthritis index, subscale pain [Mean (Standard Deviation); unit: units on a scale] — Sores of the Australian-Canadian Hand Osteoarthritis Index (AUSCAN) subscale pain ranges from 0 to 50, with higher scores indicating more pain
  units on a scale | 20.7 (11.6) | 21.7 (13.0) | 21.2 (12.3)
Australian-Canadian Hand Osteoarthritis index, subscale function [Mean (Standard Deviation); unit: units on a scale] — Scores of the Australian-Canadian Hand Osteoarthritis Index (AUSCAN) subscale function range from 0 to 90, with higher scores indicating more disability
  units on a scale | 41.3 (21.9) | 42.0 (24.9) | 41.6 (23.4)
Functional Index for Hand Osteoarthritis (FIHOA) [Mean (Standard Deviation); unit: units on a scale] — Scores of the Functional Index for Hand Osteoarthritis (FIHOA) range from 0 to 30, with higher scores indicating more disability
  units on a scale | 10.4 (0.9) | 10.3 (1.0) | 10.4 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Total Ghent University Scoring System (GUSS) of Target Joints at Week 24
Description: The Ghent University Scoring System, GUSS, is quantitative radiographic scoring system and found to be a reliable method to score radiographic change over time in erosive IP OA. It includes assessment of proportions of normal subchondral bone, subchondral plate and joint space over time. Range of score: min: 0 max:300. Change scores are measured where positive changes corresponds with remodeling or repair (better outcome), and negative changes with erosive progression (worse outcome).
Time Frame: 24 weeks
Population: intention-to-treat (ITT) population (i.e., all participants randomly assigned to groups and who attended a baseline visit)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Comparator: Experimental: Denosumab | Comparator - Placebo
Number analyzed (Participants) | 51 | 49
units on a scale | 162.2 (2.4) | 153.3 (3.2)
Statistical Analysis 1: Comparison: Active Comparator: Experimental: Denosumab vs Comparator - Placebo; Comparison between groups was done by Generalized Estimation Equations at joint level, accounting for within-patient clustering and adjusted for baseline unbalances. Missing values were imputed according to a predefined imputation model, including randomization group, baseline value and values at other time points available, presence of baseline inflammation, baseline number of affected joints; Test type: Superiority; p = 0.024, GEE; Mean Difference (Final Values) = 8.9, 95% CI 2-sided [1.0 to 16.9]

2. Secondary Outcome: Number of New Erosive Joints by Verbruggen and Veys at Week 48
Description: These are the number of new erosive IP joints according to the Verbruggen and Veys anatomical scoring system amongst the pre-erosive joints (i.e., N, S, J joints) at 48 weeks.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number; unit: joints
Units Other Than Participants: joints
Arm/Group | Active Comparator: Experimental: Denosumab | Comparator - Placebo
Number analyzed (Participants) | 46 | 46
Number analyzed (joints) | 501 | 535
joints | 9 | 38
Statistical Analysis 1: Comparison: Active Comparator: Experimental: Denosumab vs Comparator - Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.11 to 0.50]

3. Secondary Outcome: Total Ghent University Scoring System (GUSS) at Week 48
Description: The Ghent University Scoring System, GUSS, is quantitative radiographic scoring system and found to be a reliable method to score radiographic change over time in erosive IP OA. It includes assessment of proportions of normal subchondral bone, subchondral plate and joint space over time. Range of score: min: 0 max:300. Change scores are measured where positive changes corresponds with remodeling or repair, and negative changes with erosive progression.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Comparator: Experimental: Denosumab | Comparator - Placebo
Number analyzed (Participants) | 46 | 46
units on a scale | 163.5 (2.9) | 149.2 (3.9)
Statistical Analysis 1: Comparison: Active Comparator: Experimental: Denosumab vs Comparator - Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, GEE; Mean Difference (Final Values) = 14.3, 95% CI 2-sided [4.6 to 24.0]

4. Other Pre Specified Outcome: Number of (Serious) Adverse Events
Description: Number of patients who have experienced one or more (serious) adverse events throughout the study
Time Frame: 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed during the placebo controlled phase from the first dose administration up to Week 48.
Arm/Group | Active Comparator: Experimental: Denosumab | Comparator - Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 6/51 | 7/49
Other Adverse Events (participants affected / at risk) | 41/51 | 44/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Experimental: Denosumab (N=51) | Comparator - Placebo (N=49)
Major cardiovascular event (Cardiac disorders) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 3 (3)
Musculoskeletal complaints (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Infections (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Experimental: Denosumab (N=51) | Comparator - Placebo (N=49)
Infection (Infections and infestations) | 26 (41) | 22 (38)
Gastrointestinal event (Gastrointestinal disorders) | 5 (6) | 6 (7)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 5 (6)
Musculoskeletal complaints (Musculoskeletal and connective tissue disorders) | 19 (24) | 24 (34)
Nervous system disorders (incl. dizziness, vertigo, headache) (Nervous system disorders) | 4 (4) | 11 (17)
Pulmonary and respiratory complaintes (non-infectious) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rash and skin problmes (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Allergy (systemic and urticaria) (Immune system disorders) | 3 (3) | 1 (1)
Theet problems (General disorders) | 3 (3) | 3 (3)
Other (General disorders) | 4 (5) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT02771860/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT02771860/SAP_001.pdf